CLINICAL TRIAL: NCT02483585
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AMG 334 in Migraine Prevention
Brief Title: Study to Evaluate the Efficacy and Safety of Erenumab (AMG 334) Compared to Placebo in Migraine Prevention
Acronym: ARISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120297; 2014-004463-20 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-29 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Migraine
Keywords: Migraine; Headache; Episodic; Prevention; Prophylaxis
MeSH Terms: conditions — Migraine Disorders; Headache; Recurrence | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase. At week 12 participants began treatment with erenumab 70 mg administered by subcutaneous injection at weeks 12, 16, 20, 24, 28, 32, and 36 in the open-label treatment phase.
  Interventions: Drug: Placebo
- Erenumab (Experimental): Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase. Participants continued to receive erenumab 70 mg administered by subcutaneous injection at weeks 12, 16, 20, 24, 28, 32, and 36 in the open-label treatment phase.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Administered once a month by subcutaneous injection
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab
Drug: Placebo — Administered once a month by subcutaneous injection
  Arms: Placebo

SUMMARY:
To evaluate the effect of erenumab compared to placebo on the change from baseline in monthly migraine days, in adults with episodic migraine.

DETAILED DESCRIPTION:
Adults with a history of migraine with or without aura for ≥ 12 months and who experience ≥ 4 to < 15 migraine days per month with < 15 headache days per month will be randomized 1:1 to placebo or erenumab. Double-blind erenumab or placebo will be administered during the 12-week double-blind treatment phase and open-label erenumab will be administered during the 28-week open-label treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* History of migraines (with or without aura) for ≥ 12 months
* Migraine frequency: ≥ 4 and < 15 migraine days per month on average acrossthe 3 months prior to screening
* Headache (ie, migraine and non-migraine headache) frequency: < 15 headache days per month on average across the 3 months prior to screening
* Demonstrated compliance with the eDiary

Exclusion Criteria:

* Older than 50 years of age at migraine onset.
* History of cluster headache or hemiplegic migraine headache.
* Unable to differentiate migraine from other headaches
* No therapeutic response with > 2 categories for prophylactic treatment of migraine after an adequate therapeutic trial.
* Concomitant use of 2 or more medications with possible migraine prophylactic effects within 2 months prior to the start of the baseline phase or during the baseline phase. If only 1 prophylactic medication is used, the dose must be stable within 2 months prior to the start of the baseline phase and throughout the study
* Used a prohibited medication, device, or procedure within 2 months prior to the start of the baseline phase or during the baseline phase.
* Received botulinum toxin
* Anticipated to require any excluded medication, device, or procedure during the study.
* Active chronic pain syndromes (such as fibromyalgia and chronic pelvic pain).
* History of major psychiatric disorder.
* History of seizure disorder or other significant neurological conditions other than migraine.
* Human immunodeficiency virus (HIV) infection by history.
* Myocardial infarction (MI), stroke, transient ischemic attack (TIA), unstable angina, or coronary artery bypass surgery or other revascularization procedure within 12 months prior to screening.
* The subject is at risk of self-harm or harm to others. Previously randomized into an AMG 334 study.
* Unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (70):
- United States (40):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Culver City, California
  - Research Site, Long Beach, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fairfield, Connecticut
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Gurnee, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Lenexa, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Princeton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Virginia Beach, Virginia
  - Research Site, Seattle, Washington
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Glostrup Municipality
  - Research Site, Vejle
- France (4):
  - Research Site, Bordeaux
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pringy
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Portugal (3):
  - Research Site, Amadora
  - Research Site, Lisbon
  - Research Site, Torres Vedras
- Russia (4):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- Spain (7):
  - Research Site, Zaragoza, Aragon
  - Research Site, Santander, Cantabria
  - Research Site, Valladolid, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Switzerland (6):
  - Research Site, Bad Zurzach
  - Research Site, Biel
  - Research Site, Geneva
  - Research Site, Lugano
  - Research Site, Sankt Gallen
  - Research Site, Zollikon

REFERENCES:
- [Background] Dodick DW, Ashina M, Brandes JL, Kudrow D, Lanteri-Minet M, Osipova V, Palmer K, Picard H, Mikol DD, Lenz RA. ARISE: A Phase 3 randomized trial of erenumab for episodic migraine. Cephalalgia. 2018 May;38(6):1026-1037. doi: 10.1177/0333102418759786. Epub 2018 Feb 22. PMID 29471679
- [Background] Cheng S, Picard H, Zhang F, Eisele O, Mikol DD. Efficacy and safety of erenumab for migraine prevention: an overview. Japanese Journal of Headache. 2019; 45 : 493-505.
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Kawata AK, Ladd MK, Lipton RB, Buse DC, Bensink M, Shah S, Hareendran A, Mannix S, Mikol D. Reducing the physical, social, and emotional impact of episodic migraine: Results from erenumab STRIVE and ARISE phase III randomized trials. Headache. 2022 Feb;62(2):159-168. doi: 10.1111/head.14258. Epub 2022 Feb 8. PMID 35137394
- [Background] Ashina M, Kudrow D, Reuter U, Dolezil D, Silberstein S, Tepper SJ, Xue F, Picard H, Zhang F, Wang A, Zhou Y, Hong F, Klatt J, Mikol DD. Long-term tolerability and nonvascular safety of erenumab, a novel calcitonin gene-related peptide receptor antagonist for prevention of migraine: A pooled analysis of four placebo-controlled trials with long-term extensions. Cephalalgia. 2019 Dec;39(14):1798-1808. doi: 10.1177/0333102419888222. Epub 2019 Nov 10. PMID 31707815
- [Background] Kudrow D, Pascual J, Winner PK, Dodick DW, Tepper SJ, Reuter U, Hong F, Klatt J, Zhang F, Cheng S, Picard H, Eisele O, Wang J, Latham JN, Mikol DD. Vascular safety of erenumab for migraine prevention. Neurology. 2020 Feb 4;94(5):e497-e510. doi: 10.1212/WNL.0000000000008743. Epub 2019 Dec 18. PMID 31852816
- [Derived] Lampl C, Kraus V, Lehner K, Loop B, Chehrenama M, Maczynska Z, Ritter S, Klatt J, Snellman J. Safety and tolerability of erenumab in individuals with episodic or chronic migraine across age groups: a pooled analysis of placebo-controlled trials. J Headache Pain. 2022 Aug 18;23(1):104. doi: 10.1186/s10194-022-01470-4. PMID 35978286
- [Derived] Ashina M, Goadsby PJ, Dodick DW, Tepper SJ, Xue F, Zhang F, Brennan F, Paiva da Silva Lima G. Assessment of Erenumab Safety and Efficacy in Patients With Migraine With and Without Aura: A Secondary Analysis of Randomized Clinical Trials. JAMA Neurol. 2022 Feb 1;79(2):159-168. doi: 10.1001/jamaneurol.2021.4678. PMID 34928306
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 69 centers in Denmark, France, Greece, Portugal, Russia, Spain, Switzerland, and the USA. Participants were enrolled from 20 July 2015 to 19 April 2016.
Pre-assignment Details: Participants were randomized 1:1 to placebo or erenumab 70 mg once a month (QM). Randomization was stratified by region (North America vs Other) and treatment status with migraine prophylactic medication (current, prior, or no prior or current migraine prophylactic medication treatment).
Groups:
- Placebo: Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase. At week 12 participants began treatment with erenumab 70 mg administered by subcutaneous injection at weeks 12, 16, 20, 24, 28, 32, and 36 in the 28-week open-label treatment phase.
- Erenumab 70 mg QM: Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase. Participants continued to receive erenumab 70 mg administered by subcutaneous injection at weeks 12, 16, 20, 24, 28, 32, and 36 in the 28-week open-label treatment phase.
Period: Double-blind Treatment Phase
Arm/Group | Placebo | Erenumab 70 mg QM
Started | 291 | 286
Received Treatment | 289 | 283
Completed | 275 | 271
Not Completed | 16 | 15
Not completed — Decision by Sponsor | 1 | 1
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Lost to Follow-up | 3 | 2
Period: Open-label Treatment Phase
Arm/Group | Placebo | Erenumab 70 mg QM
Started | 270 (Five participants who completed the double-blind phase did not enter the open-label treatment phase) | 268 (Three participants who completed the double-blind phase did not enter the open-label treatment phase)
Completed | 243 | 243
Not Completed | 27 | 25
Not completed — Protocol-specified Criteria | 6 | 5
Not completed — Decision by Sponsor | 0 | 1
Not completed — Withdrawal by Subject | 18 | 14
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab 70 mg QM | Total
Number analyzed (Participants) | 291 | 286 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.5) | 42.3 (11.4) | 42.3 (11.4)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 290 | 283 | 573
  65 - 74 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 245 | 492
  Male | 44 | 41 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 23 | 57
  Not Hispanic or Latino | 257 | 263 | 520
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Black or African American | 27 | 24 | 51
  Multiple | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 259 | 259 | 518
  Other | 2 | 0 | 2
Region [Count of Participants; unit: Participants]
  North America | 170 | 168 | 338
  Other | 121 | 118 | 239
Treatment Status with Migraine Prophylactic Medication [Count of Participants; unit: Participants]
  Current migraine prophylactic medication treatment | 18 | 17 | 35
  Prior migraine prophylactic treatment only | 120 | 119 | 239
  No prior / current migraine prophylactic treatment | 153 | 150 | 303
Disease Duration of Migraine With or Without Aura [Mean (Standard Deviation); unit: years] | 20.03 (12.08) | 21.70 (12.62) | 20.86 (12.37)
Monthly Migraine Days [Mean (Standard Deviation); unit: days] — A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase.
  days | 8.38 (2.60) | 8.14 (2.65) | 8.26 (2.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days at Week 12
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura.
  The change from baseline in monthly migraine days was calculated as the number of migraine days during the last 4 weeks of the 12-week double-blind treatment phase - the number of migraine days during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set which includes participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in monthly migraine days in the double-blind treatment phase.
Measure: Least Squares Mean (Standard Error); unit: migraine days / month
Arm/Group | Placebo | Erenumab 70 mg QM
Number analyzed (Participants) | 288 | 282
migraine days / month | -1.84 (0.21) | -2.88 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; The primary endpoint was analyzed using a linear mixed effects model including treatment group, baseline value, stratification factors (region and prior/current treatment with migraine prophylactic medication), scheduled visit, and the interaction of treatment group with scheduled visit; Test type: Superiority — A sequential testing procedure, specifically, the hierarchical gate-keeping procedures and Hochberg method, was used to maintain the 2-sided study-wise type I error at 0.05 between the primary and efficacy secondary endpoints; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.04, 95% CI 2-sided [-1.61 to -0.47]

2. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Monthly Migraine Days at Week 12
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase and during the last 4 weeks of double-blind treatment.
  At least a 50% reduction from baseline in monthly migraine days was determined if the change in monthly migraine days from the 4-week baseline phase to the last 4 weeks of the 12-week double-blind treatment phase * 100 / baseline monthly migraine days was less than or equal to -50%.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set which includes participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in monthly migraine days in the double-blind treatment phase. Participants with missing data at week 12 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erenumab 70 mg QM
Number analyzed (Participants) | 288 | 282
percentage of participants | 29.5 | 39.7
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; Analyzed using a Cochran-Mantel-Haenszel (CMH) test after the missing data were imputed as nonresponse, stratified by stratification factors (region and prior/current treatment with migraine prophylactic medication); Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.12 to 2.27]

3. Secondary Outcome: Change From Baseline in Monthly Acute Migraine-specific Medication Treatment Days at Week 12
Description: Monthly acute migraine-specific medication treatment days is the number of days on which migraine specific medications were used between monthly doses of study drug. Migraine-specific medications includes two categories of medications: triptan-based migraine medications and ergotamine-based migraine medications.
  The change from baseline in monthly acute migraine-specific treatment days was calculated as the number of migraine-specific treatment days during the last 4 weeks of the 12-week double-blind treatment phase - the number of migraine-specific treatment days during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set which includes participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in monthly acute migraine-specific treatment days in the double-blind treatment phase.
Measure: Least Squares Mean (Standard Error); unit: acute migraine treatment days / month
Arm/Group | Placebo | Erenumab 70 mg QM
Number analyzed (Participants) | 288 | 282
acute migraine treatment days / month | -0.62 (0.14) | -1.21 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; Analyzed using a linear mixed effects model including treatment group, baseline value, stratification factors (region and prior/current treatment with migraine prophylactic medication), scheduled visit, and the interaction of treatment group with scheduled visit; Test type: Superiority; p = 0.002, Generalized Linear Mixed Model; LS Mean Difference = -0.59, 95% CI 2-sided [-0.96 to -0.21]

4. Secondary Outcome: Percentage of Participants With at Least a 5-point Reduction From Baseline in Average Impact on Everyday Activities Domain Score Measured by MPFID at Week 12
Description: The Migraine Physical Function Impact Diary (MPFID) is a self-administered 13-item instrument measuring physical functioning. It has two domains, Impact on Everyday Activities (7 items) and Physical Impairment (5 items), and one stand-alone global question. Participants completed the MPFID daily in an electronic diary based on the past 24 hours. Participants responded to each item on a 5-point scale, with difficulty items ranging from "Without any difficulty" (1) to "Unable to do" (5) and frequency items ranging from "None of the time" (1) to "All of the time" (5). For each domain, the scores were calculated as the sum of the responses and rescaled to 0 - 100, with higher scores representing greater impact of migraine.
  Achievement of at least a 5 point reduction from baseline in the monthly average domain score was calculated as (monthly average domain score during the last 4 weeks of the 12-week double-blind treatment phase - baseline monthly average domain score) was ≤ -5.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set including participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in MPFID average impact on everyday activities domain score in the double-blind treatment phase. Participants with missing post-baseline data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erenumab 70 mg QM
Number analyzed (Participants) | 288 | 282
percentage of participants | 35.8 | 40.4
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.26, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.87 to 1.71]

5. Secondary Outcome: Percentage of Participants With at Least a 5-Point Reduction From Baseline in Average Impact on Physical Impairment Domain Score Measured by MPFID at Week 12
Description: as for outcome 4
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set including participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in MPFID average impact on physical impairment domain score in the double-blind treatment phase. Participants with missing post-baseline data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erenumab 70 mg QM
Number analyzed (Participants) | 288 | 282
percentage of participants | 27.1 | 33.0
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.13, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.92 to 1.90]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4, where:
  Grade 1 = Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL); Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL; Grade 4 = Life-threatening consequences; urgent intervention indicated Grade 5 = Death related to AE.
Time Frame: From first dose of study drug up to 12 weeks after the last dose. The double-blind treatment phase was 12 weeks and the open-label treatment phase was 28 weeks.
Population: For the double-blind treatment phase adverse events were analyzed for all randomized participants who received at least one dose of study drug. For the open-label treatment phase adverse events were analyzed for all participants who received at least one dose of study drug in the open-label treatment phase.
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind Treatment Phase (12 Weeks): Placebo: Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- Double-blind Treatment Phase (12 Weeks): Erenumab 70 mg QM: Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- Open-label Treatment Phase (28 Weeks): Erenumab 70 mg QM: Participants received erenumab 70 mg administered by subcutaneous injection at weeks 12, 16, 20, 24, 28, 32, and 36 during the open-label treatment phase.
Arm/Group | Double-blind Treatment Phase (12 Weeks): Placebo | Double-blind Treatment Phase (12 Weeks): Erenumab 70 mg QM | Open-label Treatment Phase (28 Weeks): Erenumab 70 mg QM
Number analyzed (Participants) | 289 | 283 | 538
Participants
  Any adverse event | 158 | 136 | 337
  Adverse event Grade ≥ 2 | 96 | 72 | 245
  Adverse event Grade ≥ 3 | 8 | 6 | 34
  Adverse event Grade ≥ 4 | 0 | 0 | 2
  Serious adverse events | 5 | 3 | 15
  AE leading to discontinuation of study drug | 1 | 5 | 13
  Fatal adverse events | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Developed Antibodies to Erenumab
Description: Blood samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect anti-drug antibodies (ADA) against erenumab. Samples confirmed to be positive for binding antibodies were subsequently tested in a cell-based bioassay to determine neutralizing activity against erenumab (Neutralizing Antibody Assay).
  Developing antibody incidence indicates participants with a negative or no result at baseline and a positive result at any time post-baseline.
  If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the sample was defined as positive for neutralizing antibodies.
  Transient indicates a negative result at the participant's last time point tested, for those participants with a positive binding/neutralizing result post-baseline.
Time Frame: Baseline (the period prior to the first dose erenumab 70 mg) and post-baseline (the period after the first dose of erenumab 70 mg until 12 weeks after last dose, up to 48 weeks total)
Population: Participants who received at least one dose of erenumab and with post-baseline data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab 70 mg QM
Number analyzed (Participants) | 269 | 279
Participants
  Binding antibody positive | 25 | 24
  -Transient binding antibody positive | 10 | 11
  Neutralizing antibody positive | 0 | 2
  -Transient neutralizing antibody positive | 0 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 12 weeks after the last dose. The double-blind treatment phase was 12 weeks and the open-label treatment phase was 28 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Double-blind Treatment Phase (12 Weeks): Erenumab 70 mg QM: Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection the double-blind treatment phase.
Arm/Group | Double-blind Treatment Phase (12 Weeks): Placebo | Double-blind Treatment Phase (12 Weeks): Erenumab 70 mg QM | Open-label Treatment Phase (28 Weeks): Erenumab 70 mg QM
Serious Adverse Events (participants affected / at risk) | 5/289 | 3/283 | 15/538
Other Adverse Events (participants affected / at risk) | 46/289 | 54/283 | 140/538
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Phase (12 Weeks): Placebo (N=289) | Double-blind Treatment Phase (12 Weeks): Erenumab 70 mg QM (N=283) | Open-label Treatment Phase (28 Weeks): Erenumab 70 mg QM (N=538)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nasal septal operation (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Phase (12 Weeks): Placebo (N=289) | Double-blind Treatment Phase (12 Weeks): Erenumab 70 mg QM (N=283) | Open-label Treatment Phase (28 Weeks): Erenumab 70 mg QM (N=538)
Injection site pain (General disorders) | 12 | 17 | 30
Upper respiratory tract infection (Infections and infestations) | 14 | 18 | 41
Viral upper respiratory tract infection (Infections and infestations) | 17 | 17 | 53
Migraine (Nervous system disorders) | 7 | 5 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.